CLINICAL TRIAL: NCT00119457
Title: A Multi-Center, Placebo-Controlled Evaluation of the Safety and Efficacy of Three Weeks Extended VTE Prophylaxis With Daily Oral Doses of TTP889 After One Week of Standard Prophylactic Treatment Following Hip Fracture Surgery
Brief Title: Factor IX Inhibition in Thrombosis Prevention (The FIXIT Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TTP889-201; Eudract CT#2004-002511-83
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Venous Thromboembolism; Embolism and Thrombosis; Hip Fractures
Keywords: antithrombotic agents; anticoagulants; prophylaxis; embolism; deep vein thrombosis; hip fracture
MeSH Terms: conditions — Venous Thromboembolism; Embolism and Thrombosis; Hip Fractures; Embolism; Venous Thrombosis

INTERVENTIONS:
Drug: TTP889

SUMMARY:
The purpose of this study is to determine whether TTP889 prevents venous thromboembolism following surgery to repair hip fracture.

DETAILED DESCRIPTION:
FIXIT is the first Phase 2 study of TTP889. The trial is a proof-of-concept study to determine the safety and antithrombotic efficacy of TTP889 in patients at risk for venous thromboembolism (VTE). The study is a multi-center, randomized, double-blind, parallel-group evaluation of 300 mg TTP889 or placebo, administered orally once daily for three weeks, in patients who have undergone surgery to repair unilateral fracture of the upper third of either femur and who have completed 5 to 9 days of postoperative prophylactic treatment for VTE.

ELIGIBILITY:
Inclusion Criteria:

* Must have undergone reparative surgery within 72 hours after unilateral hip fracture, defined as fracture of the upper third of either femur
* Must have started standard prophylactic treatment for VTE with low molecular weight heparin (LMWH) or heparin before surgery or within 24 hours after hip fracture surgery, and continued treatment with LMWH or heparin for at least five days, but not more than nine days, after surgery
* Last dose of LMWH or heparin must have been administered at least 12 hours, but not more than 48 hours, before dosing with study drug
* Females must have a negative serum pregnancy test
* Must weigh at least 45 kg
* Must demonstrate the mental and physical ability and willingness to follow all study-specific instructions
* Must be able to read, comprehend and sign the Ethics Committee-approved informed consent form

Exclusion Criteria:

* Evidence of active bleeding
* Clinical signs of VTE
* Any medical requirement for (or intention to use) continued anticoagulation after randomization through the end of study
* History of intracranial bleeding, hemorrhagic stroke, or gastrointestinal bleeding within 3 months of study start
* Presence of active malignant disease
* Hip fracture associated with multiple trauma, that places patient at excessive risk for hemorrhage or organ system failure, or that may make it difficult or impossible to perform bilateral lower limb venography
* Intention to take aspirin at doses greater than 325 mg/day
* Hemoglobin < 5.45 mmol/L (9 g/dL), hematocrit < 29%, or a platelet count < 100,000/mL at the screening visit
* Elevated ALT or AST level > 3.0 times the ULN, or an elevated total bilirubin > 1.5 the ULN at the screening visit
* Creatinine > 180 mmol/L (2.0 mg/dL) at the screening visit
* Any other laboratory value at screening that the Investigator considers to be clinically significant and warrants exclusion from the study
* Patient is currently breast feeding a child and wishes to continue breast feeding
* Previous allergy to contrast material or any other contraindications to perform bilateral lower limb venography
* The use of another investigational drug within 28 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-01; Study Completion 2006-04

PRIMARY OUTCOMES:
To evaluate the antithrombotic efficacy of TTP889, administered once daily for three weeks, in patients who have completed standard prophylactic treatment for deep vein thrombosis after hip fracture surgery.
Evaluation of safety of once daily oral administration of TTP889 for three weeks

SECONDARY OUTCOMES:
To assess the correlation between peak and trough plasma concentrations of TTP889 and clinical safety and efficacy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt I Eriksson, MD, Study Chair — Dept of Orthopaedics, Goteborg University; David P Ward, MD, Study Director — vTv Therapeutics
Locations (21):
- Czechia (5):
  - Nemocnice Ceske Budejovice, Urazove oddeleni, České Budějovice
  - FN s Poliklinikou Ostrava, Traumatologicke Centrum, Ostrava-Poruba
  - FN Motol, Ortopedicka Klinicka UK 2.LF a FN Notol, Prague
  - FN Na Bulovce, Ortopedicka Klinika IPVZ a 1.LF UK ORT, Budinova 2, Prague
  - VFN, I. Chirurgicka klinika, Praha-2
- Denmark (7):
  - AAlborg Hospital, Aalborg
  - H:S Bispebjerg Hospital, Copenhagen
  - Ortopaedkirurgisk Klinik, Farso, Farsø
  - Amtsygehuset i Gentofte, Hellerup
  - KAS Herlev, Herlev
  - Horsholm Hospital, Hørsholm
  - Silkeborg Hospital, Silkeborg
- Norway (4):
  - Orthopedics, Alesund Sykehus, Ålesund
  - Skyehuset Innlandet HF, Gjøvik
  - Skyehuset Innlandet HF, Lillehammer
  - Halfdan Wilhelmsens Alle 17, Tønsberg
- Sweden (5):
  - Ortoped Kliniken, Sahlgrenska Universitetssjukhus, Ostra, Gothenburg
  - Ortopedsektionen, Kirurgkliniken, Kungalvs Sjukhus, Kungälv
  - Ortoped kliniken, Sahlgrenska Universitetssjukhus, Mölndal
  - Ortoped kliniken, NU-sjukvarden, Udevalla Sjukhus, Udevalla
  - Ortoped kliniken, Sjukhuset i Varberg, Varberg

REFERENCES:
- [Derived] Eriksson BI, Dahl OE, Lassen MR, Ward DP, Rothlein R, Davis G, Turpie AG; Fixit Study Group. Partial factor IXa inhibition with TTP889 for prevention of venous thromboembolism: an exploratory study. J Thromb Haemost. 2008 Mar;6(3):457-63. doi: 10.1111/j.1538-7836.2007.02872.x. Epub 2007 Dec 12. PMID 18088349